CLINICAL TRIAL: NCT05167890
Title: Impact of Standardized Coffee Versus Orange Juice Intake on Enhancing Bowel Movements After Elective Laparoscopic Colorectal Surgery, RCT
Brief Title: Impact of Coffee vs Orange Juice on Enhancing Recovery After Laparoscopic Colorectal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Yasser Debakey, Lecturer of surgical oncology, NCI, Cairo University, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Debakey2
Record Dates: First submitted 2021-11-30; First posted 2021-12-22 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Colorectal Surgery
MeSH Terms: interventions — Coffee

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coffee Arm (Active Comparator): Patients in coffee arm receive 1 cup of coffee 3 times per day (150 mL at 8:00 AM, 12:00 PM, and5:00 PM), in addition to the regular infusion therapy and/or alimentation starting the first day postoperatively till the end of the 3 postoperative day.
  Interventions: Dietary Supplement: Coffee
- Orange Arm (Active Comparator): Patients in orange arm receive 1 cup of orange juice 3 times per day (150 mL at 8:00 AM, 12:00 PM, and5:00 PM), in addition to the regular infusion therapy and/or alimentation starting the first day postoperatively till the end of the 3 postoperative day.
  Interventions: Dietary Supplement: Orange juice

INTERVENTIONS:
Dietary Supplement: Coffee — Coffee 3 times per day
  Arms: Coffee Arm
Dietary Supplement: Orange juice — Orange juice 3 times per day
  Arms: Orange Arm

SUMMARY:
Colorectal surgery, even performed by laparoscopy is followed by a transient episode of GI hypomotility, which results in a postoperative ileus (POI). The usual duration of this benign postoperative situation varies between 3 and 5 days for colon surgery. A longer duration of POI will result in more postoperative complications such as delayed surgical wound healing, atelectasis, pneumonia, and deep vein thrombosis; in a prolonged hospital stay; and increased healthcare cost. Different studies reported that the duration of POI correlates with total surgery time, blood loss, total opiate dose degree of surgical trauma, and bowel manipulation. Many attempts have been made to reduce the phase of postoperative intestinal hypomotility. The different strategies are well described in enhanced recovery and fast-track concepts and focus on minimal surgical trauma, rapid postoperative mobilization, early feeding, preemotive laxative treatment, restrictive fluid management, and minimal postoperative opioid prescription. Furthermore, several pharmacologic agents have been evaluated; however, not all offered a convincing benefit, nor were they free of adverse effects. Coffee is a worldwide highly consumed beverage, offering pleasure to many people of different cultures, and which many associate with an increase of bowel function.

The aim of this study is to compare the time to first bowel movement after laparoscopic colorectal surgery between patients drinking coffee or orange juice postoperatively, in a randomized controlled trial (RCT).

DETAILED DESCRIPTION:
The study is designed as a multi-center, open-label RCT. All of the eligible patients undergoing elective laparoscopic colon or rectal resection are considered for participation in the study unless exclusion criteria are present. Written informed consent is obtained after hospital admission.

Patients will be classified into two groups:

1. Coffee Arm: receiving coffee (Turkish sugar free coffee).
2. Orange Arm: receiving orange juice (fresh sugar free). Baseline demographics, peri-operative data (HB, serum Alb and electrolytes), duration of operation, conversion rate to open surgery, estimated blood loss, short-term outcome, and LOS (length of hospital stay) will be analyzed.

Exclusion criteria:

Creation of a colostomy or ileostomy, Any additional small bowel anastomosis, Emergency operations, known hypersensitivity or allergy to coffee or orange.

Patients in coffee arm receive 1 cup of coffee 3 times per day (150 mL at 8:00 AM, 12:00 PM, and5:00 PM), in addition to the regular infusion therapy and/or alimentation starting the first day postoperatively till the end of the 3 postoperative day. In orange arm, the same protocol is applied, replacing coffee with orange juice. All of the patients drink the same quantity of each drink.

Methodology Type of study: open-labeled randomized controlled trial The assignment of patients to either group will be done by a random computer-assissted allocation. The allocation will be done by the use of opaque envelopes with assignments.

Follow up: will be completed within one month (immediate post-operative outcome).

Outcome Measures:

* primary end point was time to first bowel movement (flatus or stool) starting at the time of surgery completion. Included patients are given a diary and are asked (after instruction) to document on a daily basis if they had defecation or flatus and what time; this was verified 3 times per day by the nurse.
* Secondary end points include the number of postoperative bowel movements until discharge, length of hospital stay, and postoperative complications (Dindo-Clavien classification) and are documented by the resident in charge of the patient. All of the patients are discharged with an appointment for a 30-day follow-up

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective laparoscopic colon or rectal resection

Exclusion Criteria:

* Creation of a colostomy or ileostomy,
* Any additional small bowel anastomosis,
* Emergency operations,
* known hypersensitivity or allergy to coffee or orange.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-11-22 (Actual); Primary Completion 2023-01-22 (Estimated); Study Completion 2023-01-25 (Estimated)

PRIMARY OUTCOMES:
Primary end point is time to first bowel movement (flatus or stool) starting at the time of surgery completion. | From day of surgery to-day of hospital discharge (up to 2 weeks)
  Included patients are given a diary and are asked (after instruction) to document on a daily basis if they had defecation or flatus and what time; this was verified 3 times per day by the nurse.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Mahmoud, Professor, Study Director — National Cancer Institute, Cairo University, Egypt
Locations (1):
- National Cancer Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
In a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publication and for a year
Access Criteria: The journal of publication